CLINICAL TRIAL: NCT07177703
Title: A Prospective Single-arm Exploratory Study on the Efficacy and Safety of Treprostinil Injection in the Treatment of Patients With Intermediate-risk Pulmonary Arterial Hypertension
Brief Title: Efficacy and Safety of Treprostinil in Intermediate-Risk Pulmonary Arterial Hypertension
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Junbo Ge, Director of Cardiology, Shanghai Zhongshan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tre-ImPAH
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Arterial Hypertension (PAH)
Keywords: PAH; Treprostinil
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Treatment is added to the participant's stable background regimen of standard-of-care oral PAH therapies (e.g., endothelin receptor antagonists, phosphodiesterase-5 inhibitors, and/or soluble guanylate cyclase stimulators).
  Treprostinil is initiated at a dose of 1.25 ng/kg/min. The dose is then titrated upwards based on individual patient tolerability and clinical response. The planned titration schedule is an increase of 1.25 ng/kg/min weekly for the first four weeks of treatment, followed by weekly increases of 2.5 ng/kg/min thereafter, as tolerated.
  Interventions: Drug: Treprostinil

INTERVENTIONS:
Drug: Treprostinil — Treprostinil is initiated at a dose of 1.25 ng/kg/min. The dose is then titrated upwards based on individual patient tolerability and clinical response. The planned titration schedule is an increase of 1.25 ng/kg/min weekly for the first four weeks of treatment, followed by weekly increases of 2.5 ng/kg/min thereafter, as tolerated.

SUMMARY:
Pulmonary Arterial Hypertension (PAH) is a serious condition that puts strain on the right side of the heart. While oral medications can help, many patients with intermediate-risk PAH may not see enough improvement, and their heart function can continue to decline.

This study aims to find out if adding an injectable medication, Treprostinil, to a patient's current oral PAH therapy can improve heart function and overall health. This is a single-arm study, which means all participants will receive the study treatment.

The main goal is to measure the change in the amount of blood the right side of the heart pumps with each beat (Right Ventricular Stroke Volume, or RVSV) after 3 months of treatment. This will be measured using a specialized heart scan called Cardiac Magnetic Resonance Imaging (CMR). Researchers will also assess changes in exercise ability (with a 6-minute walk test), blood markers, and patient symptoms.

Participants will be in the main part of the study for 3 months, with follow-up for a total of 24 months to monitor the long-term effects and safety of the treatment.

DETAILED DESCRIPTION:
Background and Rationale:

Pulmonary Arterial Hypertension (PAH) is a progressive vasculopathy leading to increased pulmonary vascular resistance, right ventricular (RV) failure, and mortality. While guidelines recommend initial combination oral therapy, a substantial number of patients, particularly those at intermediate-risk, do not achieve a low-risk status. Subclinical RV deterioration can occur even in seemingly stable patients, suggesting that more intensive therapeutic strategies may be warranted to improve long-term outcomes.

Parenteral prostacyclin analogues, like Treprostinil, are potent therapies recommended for high-risk PAH. However, there is a lack of prospective data on their efficacy in inducing positive RV remodeling and improving clinical outcomes when initiated in patients with intermediate-risk PAH who are already on background oral therapies. This study aims to address this evidence gap.

Study Design and Objectives:

This is a prospective, single-center, single-arm, open-label, exploratory study designed to evaluate the efficacy and safety of adding subcutaneous Treprostinil to standard-of-care oral therapy for patients with intermediate-risk PAH.

The primary objective is to assess the change from baseline in Right Ventricular Stroke Volume (RVSV) at 3 months, as measured by Cardiac Magnetic Resonance (CMR). The hypothesis is that the addition of Treprostinil will lead to a significant improvement in RVSV, reflecting favorable RV remodeling.

Secondary objectives include evaluating changes from baseline in:

WHO Functional Class (FC) 6-minute walk distance (6MWD) N-terminal pro-B-type natriuretic peptide (NT-proBNP) levels Other CMR-derived parameters of RV structure and function (e.g., RV ejection fraction [RVEF], RV end-systolic volume index [RVESVI]) Risk stratification scores Incidence of clinical worsening events over the follow-up period. Exploratory objectives include the assessment of changes in other echocardiographic parameters, health-related quality of life, and a panel of serum biomarkers associated with inflammation and cardiac remodeling (e.g., TNF-α, IL-6, MMP2, TIMP1).

Methodology:

A total of 32 eligible patients with intermediate-risk PAH will be enrolled. Participants must be on a stable dose of at least one oral PAH-targeted therapy (e.g., an endothelin receptor antagonist and/or a phosphodiesterase-5 inhibitor/soluble guanylate cyclase stimulator) or be treatment-naïve and willing to start oral therapy concurrently.

All participants will initiate subcutaneous Treprostinil, with the dose titrated according to tolerability and clinical response, following the product's prescribing information.

Comprehensive assessments, including CMR, 6MWD, WHO FC, and laboratory tests, will be performed at baseline and at 3 months. Further follow-up assessments will occur at 1 month and continue for a total of 24 months to evaluate long-term safety and outcomes. Safety will be monitored throughout the study by recording all adverse events and laboratory abnormalities.

ELIGIBILITY:
Inclusion Criteria:

* Signed the informed consent form.
* Age between 18 and 75 years, inclusive.
* Diagnosed with Pulmonary Arterial Hypertension (PAH, WHO Group 1) of the following etiologies:Idiopathic;Heritable;Drug or toxin-induced (excluding amphetamine-induced PAH);Associated with repaired congenital systemic-to-pulmonary shunts (repair performed ≥1 year prior);Associated with connective tissue disease;Associated with HIV infection;
* Has undergone a right heart catheterization (RHC) within 6 months of the baseline visit.
* Baseline RHC demonstrates the following hemodynamics:Mean pulmonary arterial pressure (mPAP) > 20 mmHg;Pulmonary artery wedge pressure (PAWP) ≤ 15 mmHg;Pulmonary vascular resistance (PVR) > 2 Wood units;
* WHO Functional Class II, III, or IV.
* Risk stratification according to 2022 ESC/ERS guidelines is either intermediate-risk at initial diagnosis or low- to intermediate-risk during follow-up.
* Patient is on a stable dose of an endothelin receptor antagonist (ERA) and/or a phosphodiesterase-5 inhibitor (PDE-5i) or a soluble guanylate cyclase (sGC) stimulator for at least 30 days prior to baseline; OR, if treatment-naïve, is willing to initiate one of these therapies in addition to the study drug.

Exclusion Criteria:

* Age < 18 years.
* Diagnosis of Pulmonary Hypertension belonging to WHO Groups 2, 3, 4, or 5.
* Patients undergoing dialysis.
* Severe hepatic impairment (Child-Pugh Class C).
* Use of any prostacyclin-pathway drugs (epoprostenol, treprostinil, iloprost, beraprost, or selexipag) within 30 days prior to the baseline visit.
* Presence of implanted metallic devices that would interfere with Cardiac - - - Magnetic Resonance (CMR) imaging, such as defibrillators, neurostimulators, cochlear implants, permanent infusion devices, implanted pumps, or certain plates/screws.
* In the investigator's judgment, the patient is unable to complete or comply with study requirements.
* Refusal to sign the informed consent form or refusal to participate in follow-up visits.
* Participation in any other clinical trial involving an investigational drug, device, or procedure within 30 days prior to the baseline visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-10-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Right Ventricular Stroke Volume (RVSV) | 3 months
  Change in Right Ventricular Stroke Volume (RVSV) from baseline, as measured by Cardiac Magnetic Resonance (CMR). RVSV is the volume of blood pumped from the right ventricle of the heart during one contraction.

IPD SHARING:
Plan to Share IPD: Undecided